CLINICAL TRIAL: NCT07175961
Title: Improving Survivorship for Critically Ill Patients Aged 65 and Over
Acronym: IMPROVE-65
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ANZIC-RC/CH007
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Recovery Outcomes; Care Coordination
Keywords: critical illness; recovery coordination; patient reported outcomes
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Standard care (No Intervention): Paticipants randomised to the control group will not receive the intervention. They will be contacted by the study team to collect data on access to primary health care services post hospital discharge and will be contacted at D90 and D180 by outcome assessors to collected patient reported outcomes.
- Intervention (Experimental): Participants randomised into this group will receive tailored care coordination and support to develop recovery goals post hospital discharge.
  Interventions: Other: Multicomponent telehealth care coordination

INTERVENTIONS:
Other: Multicomponent telehealth care coordination — Participants randomised into the intervention group will be assigned a recovery navigator prior to discharge from hospital. The recovery navigator will provide the participant with a study tailored discharge summary, arrange the patients first appointment with their general practitioner and will ensure medications are reconciled prior to hospital discharge. The recovery coordinator will arrange weekly calls with the participant for the first 4 weeks and then fortnightly until week 12 to set recovery goals and assess recovery goals and navigator further primary care support if required. Participants will also be called at Day 90 and 180 by outcome assessors to collected patient reported outcomes.
  Arms: Intervention

SUMMARY:
IMPROVE-65 is a randomised control trial designed specifically for people aged over 65 who have survived critical illness. It aims to support patients and general practitioners by providing timely, personalised information to help them work together to make informed goals and decisions about their care after hospital discharge. The aim of the study is to improve recovery and avoid preventable hospital readmissions.

DETAILED DESCRIPTION:
Critical illness and intensive care unit (ICU) admissions represent significant life events that carry substantial risks for long-term health consequences. An estimated 50% of Australians will be admitted to ICU during their lifetime, placing them at considerable risk of new or worsened physical, cognitive, and psychological dysfunction following discharge. Among ICU patients, those aged 65 years and older constitute the majority, accounting for 52.5% of all admissions. Older adults experience disproportionately higher burdens of illness severity, frailty, and comorbidities, which complicate both the management of acute critical illness and the subsequent recovery process. These factors contribute to longer ICU and hospital stays, increased mortality, and a heightened risk of long-term disability. Previous research shows that nearly 40% of Australian ICU patients aged over 65 years are living with significant disability six months after discharge.

Despite the growing number of ICU survivors and the known risks of long-term morbidity, there is currently no formal or standardised system of follow-up care in Australia to monitor or support recovery. Survivors of critical illness have frequently reported fragmented transitions from hospital to home, poor communication between tertiary and primary care providers, and insufficient support to prevent or manage new disability. General practitioners (GPs), often the primary source of ongoing care, have similarly identified a lack of communication and the absence of prioritised discharge summaries as barriers to effective post-ICU care.

Building on these insights, previous work has explored innovative models of care to support functional recovery. This includes care navigation to reduce avoidable hospitalisations among high-risk patients, digital tools to improve communication between hospital and primary care, and technology-enabled goal-setting to facilitate rehabilitation. These initiatives demonstrate the potential for digital and telehealth approaches to bridge existing gaps in care continuity and patient-centred recovery.

This trial will determine if a multifaceted recovery navigated approach to coordinate and deliver timely and individualised post hospital care and recovery goals, will reduce the burden of new disability at 3 months following discharge from hospital after critical illness. Additionally, the trial will review the cost effectiveness at 6 months after randomisation. By enabling more effective communication between ICU survivors and their GPs, improving access to health information, and promoting shared decision-making, IMPROVE-65 aims to enhance the quality of survivorship, reduce new disability, and minimise healthcare costs and avoidable hospital readmissions for critically ill older adults.

ELIGIBILITY:
Inclusion Criteria:

* Was admitted to ICU for at least 48 hours
* is aged 65 years or older at the time of hospital admission
* Is alive and ready for hospital discharge
* Is expected to survive for 6 months beyond hospital discharge (e.g. not discharged on palliative care)
* Has new disability at hospital discharge measured using the global disability scale

Exclusion Criteria:

* Is not expected to reside in Australia for 3 months following randomisation.
* Is not expected to be living at home within 2 weeks of acute hospital discharge (e.g. prolonged inpatient rehabilitation)
* Is unable to identify a GP or GP clinic and/or are unable or unwilling to attend a GP appointment scheduled by the recovery navigator.
* Has an existing recovery or nurse navigator as part of their routine clinical care to assist with planning their care after hospital discharge

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite endpoint of death, avoidable hospital readmission and new global disability measured using the World Health Organisation Disability Schedule (WHODAS) 2.0 12L at 90 days after randomisation. | From randomisation until 90 days post randomisation.
  The hierarchical outcome of interest is a combination of out-of-hospital mortality, need for hospital readmission and WHODAS 2.0 score. The primary composite endpoint will be analysed using the win odds to account for ties.

SECONDARY OUTCOMES:
All-cause mortality to day 180 | From randomisation until Day 180 outcome assessment is completed.
Avoidable acute hospital readmissions to day 90 | From randomisation until day 90 post randomisation
  Measured by reviewing the number of emergency admissions to hospital participants had between randomisation and day 90.
Patient Activation Measure (PAM) at day 90 | From randomisation until Day 90 post randomisation.
Activities of Daily Living at Day 90 | From randomisation until Day 90 outcome assessment is completed.
  Measured with the EuroQoL 5-Dimension, 5-Level (EQ-5D-5L). Five questions are asked relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has five response options from 1 (no problems) to 5 (extreme problems).
Self-rated health at Day 90 | From randomisation until Day 90
  Measured using the EQ-Visual Analogue Scale (EQ-VAS) at Day 180. Measured on a scale of 0 to 100. The participant is asked to rate their health on the day of the assessment with 0 being the worst health and 100 being the best.
Activities of Daily Living at Day 180 | From randomisation until Day 180
  Measured with the EuroQoL 5-Dimension, 5-Level (EQ-5D-5L). Five questions are asked relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has five response options from 1 (no problems) to 5 (extreme problems).
Self-rated health at Day 180 | From randomisation to Day 180
  Measured using the EQ-Visual Analogue Scale (EQ-VAS) at Day 180. Measured on a scale of 0 to 100. The participant is asked to rate their health on the day of the assessment with 0 being the worst health and 100 being the best.
New disability at Day 90 | From randomisation to Day 90 outcome assessment is completed.
  Measured with the World Health Organization Disability Assessment Schedule 2.0 Proxy Administered. (WHODAS 2.0 12L). New disability is considered a change in WHODAS >10% from baseline). The participant is asked 12 questions relating to cognition, mobility, self-care, interacting with people, life activities and participation. Each question is ranked on a 5-point Likert scale from 0 (None) to 4 (Extreme or cannot do). The total score is the sum of all 12 question and can range from 0 to 48 with a higher score indicating a greater degree of disability or function.
New disability at Day 180 | From randomisation until Day 180 assessment is complete
  Measured with the World Health Organization Disability Assessment Schedule 2.0 Proxy Administered. (WHODAS 2.0 12L). New disability is considered a change in WHODAS >10% from baseline). The participant is asked 12 questions relating to cognition, mobility, self-care, interacting with people, life activities and participation. Each question is ranked on a 5-point Likert scale from 0 (None) to 4 (Extreme or cannot do). The total score is the sum of all 12 question and can range from 0 to 48 with a higher score indicating a greater degree of disability or function.
Activities of daily living at day 90 | From randomisation until Day 90
  Measured using the Katz Index of Independence in Activities of Daily Living (ADL) which assesses basic activities of daily living. The participant is asked about 6 categories of daily living and given a score of 0 or 1 based on their ability to complete the task either independently or with support. A final score between 0 and 6 is calculated, with the higher score indicating greater independence.
Activities of daily living at day 180 | From randomisation until day 180
  Measured using the Katz Index of Independence in Activities of Daily Living (ADL) which assesses basic activities of daily living. The participant is asked about 6 categories of daily living and given a score of 0 or 1 based on their ability to complete the task either independently or with support. A final score between 0 and 6 is calculated, with the higher score indicating greater independence.
Instrumental activities of daily living at day 90 | From randomisation until day 90
  Measured using the Lawton Instrumental Activities of Daily Living Scale. Eight categories of daily activities are asked, and the participant is scored for each category with either a 0 or a 1 based on the highest functional level for each activity. The overall score will be between 0 and 8 with higher scores indicating greater functional independence.
Instrumental activities of daily living at day 180 | From randomisation until day 180
  Measured using the Lawton Instrumental Activities of Daily Living Scale. Eight categories of daily activities are asked, and the participant is scored for each category with either a 0 or a 1 based on the highest functional level for each activity. The overall score will be between 0 and 8 with higher scores indicating greater functional independence.
Anxiety and Depression at day 180 | From randomisation until Day 180 outcome assessment is completed.
  Measured using the Hospital Anxiety and Depression scale (HADs) which is a 14 item scale that consists of two seven item sub-scales; seven questions for anxiety and seven questions for depression. The scale is measured with each item measured on a four point Likert scale (0 to 3). The higher the score indicating the greater the severity.
Participant cognition at day 180 | At day 180 from randomisation
  Measured using the Montreal Cognitive Assessment Blind (MOCA-Blind)
Post traumatic stress disorder at day 180 | Measured at Day 180 after randomisation
  Measured using the Impact of Events Scale 6 Items that consists of 6 questions all measured on a 5-point Likert scale from 0 to 4 with the higher the score indicating greater severity.
  0 - Not at all; 1 - A little bit; 2 - Moderately; 3 - Quite a bit; 4 - Extremely
Cost-effectiveness of the intervention at day 180 | From randomisation until Day 180.
  The primary cost-effectiveness analysis will be conducted from the Australian healthcare payer's perspective using an analytical time horizon of 6-months. Post discharge costs will be determined using patient-level data linkage to determine long-term health care use (including readmission to hospital and emergency department presentation). Quality-adjusted life years (QALYs) will be calculated using information from the Euroqol 5-dimension 5 level (EQ-5D-5L) assessed at day 180 post randomisation, combined with information on vital status. We will calculate incremental cost-effectiveness ratios, including the cost per additional QALY for the intervention versus standard care. To increase the robustness of the sampling, we will use non-parametric bootstrapping with unrestricted random sampling to produce cost and effectiveness replications, and confidence intervals for the cost-effectiveness ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, Professor, Study Chair — Monash University
Locations (2):
- Australia (2):
  - Cabrini Hospital Malvern, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, the study management committee will consider requests from researchers who provide a methodologically sound scientific proposal as per the Data Sharing Policy set out in the ANZIC Research Centre Terms of Reference.